CLINICAL TRIAL: NCT03574558
Title: Personalized Automated Determination of Insulin Pump Setting for Subjects With Type 1 Diabetes Switching From MDI to Pump Therapy and Vice Versa- Safety and Efficacy Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Jaeb Center for Health Research (Other); DreaMed (Industry); University of Padova (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC0409-18ctil
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-01

CONDITIONS: Type1diabetes
Keywords: Pump therapy; Multiple Daily Injections (MDI); Decision Support System (DSS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MD-Logic Switch Advisor (Experimental): MD-Logic Switch Advisor Algorithm for personalized automated determination of insulin pump settings for subjects with type 1 diabetes switching from MDI to pump therapy and vice versa
  Interventions: Device: MD-Logic Switch Advisor

INTERVENTIONS:
Device: MD-Logic Switch Advisor — Study algorithm will be used in order to determine the initial pump setting/ MDI dosing while switching from from MDI to pump therapy or vice versa

SUMMARY:
The "MD-Logic Switch Advisor" is a software product that is designed to assist in insulin dosage decision making and has two components:

A. MD-Logic Switch Advisor for initiation of pump therapy - this product is designed to assist physicians in decision making when initiating insulin pump therapy.

B. MD-Logic Switch Advisor for patients who use insulin pump therapy and need to switch to MDI (Multiple Daily Injections).

This feasibility study will be divided to two parts:

part A - will include up to 20 patients to evaluate in a feasibility study the switch Advisor from MDI to pump therapy part B - will include up to 20 patients to evaluate in a feasibility study the switch Advisor from pump therapy to MDI The main objective is to evaluate the safety and efficacy of using the MD-Logic Switch Advisor to determine insulin dosing for subjects with type 1 diabetes using pump therapy who wish to switch to from pump to MDI therapy and vice versa.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has documented Type 1 Diabetes Mellitus, as defined by the American Diabetes Association and World Health Organization (ADA/WHO) for at least 3 months prior to study enrolment ( Part A of the study) or at least 6 months (Part B of the study)
2. Insulin dose requirement is equal or above 0.5/unit/kg
3. The subject age is ≥ 6 years and below 30 years at the time of enrolment
4. A1c < 10%
5. The subject uses multiple daily injections to deliver insulin and wish to switch to pump therapy (Part A of the study) or the subject uses pump therapy for at least 3 months and is willing to switch to multiple daily injections for the study period (Part B of the study)
6. The subject is willing to follow study instructions
7. Subject is available for entire study duration

Exclusion Criteria:

1. Any significant diseases / conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study or compromise patient's safety, or that influence metabolic control (e.g. anemia, significantly impaired hepatic function, renal failure, history of adrenal insufficiency).
2. Subject is taking or has taken oral or parenteral glucocorticoids within 1 month prior to screening or plans to take oral or parenteral glucocorticoids within the planned study duration. Exceptions: Short term oral or paraenteral glucocorticoids up to 7 days
3. Subject has known allergy to medical grade adhesives
4. Subject is participating in another study of a medical device or drug that could affect glucose measurements or glucose management or receipt of any investigational medical product within 1 month prior to screening (visit1)
5. Female subject of child-bearing potential who have a positive pregnancy test at screening, is pregnant, breast-feeding, or planning to become pregnant within the planned study duration (or is not using adequate contraceptive methods)
6. Subject diagnosed with current eating disorder such as anorexia or bulimia
7. Subject has a history of one or more episodes of Diabetes Keto-acidosis requiring hospitalization within a 3 months prior to screening
8. Subject has visual impairment or hearing loss, which in the Investigator's opinion, may compromise patient ability to perform study procedures safely (child and parent should be evaluated as a unit)

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Number of hypoglycemic below 54 mg/dl | Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Schnider children's medical center, Petah Tikva, Israel